CLINICAL TRIAL: NCT00843271
Title: Endothelial Dysfunction, Biomarkers, and Lung Function (MESA LUNG)
Brief Title: Endothelial Dysfunction, Biomarkers, and Lung Function -Ancillary to MESA
Acronym: MESA-LUNG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAA7791; R01HL077612 (NIH); NCT00094224 (obsolete NCT alias)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Emphysema; Endothelial Dysfunction
Keywords: COPD MESA LUNG BIOMARKERS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MESA Lung: MESA-Lung is an ancillary study of the Multi-Ethnic Study of Atherosclerosis (MESA). MESA, established in 1999, is well characterized, multi-ethnic (white, Black, Hispanic and Chinese), and multi-center (Columbia, Johns Hopkins, Northwestern, UCLA, Minnesota,and Wake Forest) prospective cohort study. MESA-Lung included a 60% random sample of the MESA cohort at the six Field Centers in Exam 3 and Exam 4, stratified on race/ethnicity.

SUMMARY:
The purpose of MESA-Lung is to assess the role of endothelial dysfunction and genetic susceptibility in subclinical COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is currently the fourth leading cause of death in the United States, and morbidity and mortality from COPD continue to rise. Despite the magnitude of the problem, therapeutic options are limited - particularly in comparison to cardiovascular disease. Smoking cessation is essential to the treatment and prevention of COPD. However, although smoking is the principal cause of COPD, only a minority of smokers develops symptomatic COPD and many former smokers develop COPD years to decades after they have stopped smoking. The only other medical intervention proven to reduce mortality from COPD is supplemental oxygen therapy. There is therefore an urgent need for newer understandings of the pathophysiology of COPD that might lead to the development of better therapies for COPD.

MESA-Lung is ancillary of the ongoing Multi-Ethnic Study of Atherosclerosis (MESA). MESA-lung will utilize the various existing measures of endothelial function that have been already been collected in MESA (flow-mediated dilatation [FMD] and related biomarkers and gene polymorphisms) to test the hypotheses that the endothelial dysfunction occurs in the clinical COPD.

ELIGIBILITY:
Inclusion Criteria:

* A random sample of MESA participants active at Exam 3 and/or 4.

Exclusion Criteria:

* MESA participants without MESA Exam 3 or 4 measurements.
* MESA participants without FMD measurements in Exam 1.
* MESA participants who have not consented to genetic testing.

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MESA cohort
Sampling Method: Non-Probability Sample
Enrollment: 4359 (Actual)
Dates: Start 2004-10; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Lung Function | 2004-2011

SECONDARY OUTCOMES:
Lung Density | 2000-2011

CONTACTS AND LOCATIONS:
Overall Officials: R. Graham Barr, M.D., Dr.PH., Principal Investigator — Columbia University

REFERENCES:
- [Result] He K, Liu K, Daviglus ML, Mayer-Davis E, Jenny NS, Jiang R, Ouyang P, Steffen LM, Siscovick D, Wu C, Barr RG, Tsai M, Burke GL. Intakes of long-chain n-3 polyunsaturated fatty acids and fish in relation to measurements of subclinical atherosclerosis. Am J Clin Nutr. 2008 Oct;88(4):1111-8. doi: 10.1093/ajcn/88.4.1111. PMID 18842801
- [Result] Jiang R, Burke GL, Enright PL, Newman AB, Margolis HG, Cushman M, Tracy RP, Wang Y, Kronmal RA, Barr RG. Inflammatory markers and longitudinal lung function decline in the elderly. Am J Epidemiol. 2008 Sep 15;168(6):602-10. doi: 10.1093/aje/kwn174. Epub 2008 Aug 6. PMID 18687665
- [Result] Mesia-Vela S, Yeh CC, Austin JH, Dounel M, Powell CA, Reeves A, Santella RM, Stevenson L, Yankelevitz D, Barr RG. Plasma carbonyls do not correlate with lung function or computed tomography measures of lung density in older smokers. Biomarkers. 2008 Jun;13(4):422-34. doi: 10.1080/13547500802002859. PMID 18484356
- [Result] Jiang R, Camargo CA Jr, Varraso R, Paik DC, Willett WC, Barr RG. Consumption of cured meats and prospective risk of chronic obstructive pulmonary disease in women. Am J Clin Nutr. 2008 Apr;87(4):1002-8. doi: 10.1093/ajcn/87.4.1002. PMID 18400725
- [Result] Barr RG, Stemple KJ, Mesia-Vela S, Basner RC, Derk SJ, Henneberger PK, Milton DK, Taveras B. Reproducibility and validity of a handheld spirometer. Respir Care. 2008 Apr;53(4):433-41. PMID 18364054
- [Result] Arehart E, Stitham J, Asselbergs FW, Douville K, MacKenzie T, Fetalvero KM, Gleim S, Kasza Z, Rao Y, Martel L, Segel S, Robb J, Kaplan A, Simons M, Powell RJ, Moore JH, Rimm EB, Martin KA, Hwa J. Acceleration of cardiovascular disease by a dysfunctional prostacyclin receptor mutation: potential implications for cyclooxygenase-2 inhibition. Circ Res. 2008 Apr 25;102(8):986-93. doi: 10.1161/CIRCRESAHA.107.165936. Epub 2008 Mar 6. PMID 18323528
- [Result] Lederer DJ, Benn EK, Barr RG, Wilt JS, Reilly G, Sonett JR, Arcasoy SM, Kawut SM. Racial differences in waiting list outcomes in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Feb 15;177(4):450-4. doi: 10.1164/rccm.200708-1260OC. Epub 2007 Nov 15. PMID 18006881
- [Result] Barr RG, Mesia-Vela S, Austin JH, Basner RC, Keller BM, Reeves AP, Shimbo D, Stevenson L. Impaired flow-mediated dilation is associated with low pulmonary function and emphysema in ex-smokers: the Emphysema and Cancer Action Project (EMCAP) Study. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1200-7. doi: 10.1164/rccm.200707-980OC. Epub 2007 Aug 29. PMID 17761614
- [Result] Varraso R, Fung TT, Barr RG, Hu FB, Willett W, Camargo CA Jr. Prospective study of dietary patterns and chronic obstructive pulmonary disease among US women. Am J Clin Nutr. 2007 Aug;86(2):488-95. doi: 10.1093/ajcn/86.2.488. PMID 17684223
- [Result] Jones DP, Camargo CA Jr, Speizer FE, Barr RG. Prospective study of short stature and newly diagnosed asthma in women. J Asthma. 2007 May;44(4):291-5. doi: 10.1080/02770900701344116. PMID 17530528
- [Result] Jiang R, Paik DC, Hankinson JL, Barr RG. Cured meat consumption, lung function, and chronic obstructive pulmonary disease among United States adults. Am J Respir Crit Care Med. 2007 Apr 15;175(8):798-804. doi: 10.1164/rccm.200607-969OC. Epub 2007 Jan 25. PMID 17255565
- [Result] Barr RG, Bourbeau J, Camargo CA, Ram FS. Tiotropium for stable chronic obstructive pulmonary disease: A meta-analysis. Thorax. 2006 Oct;61(10):854-62. doi: 10.1136/thx.2006.063271. Epub 2006 Jul 14. PMID 16844726
- [Result] Jiang R, Jacobs DR Jr, Mayer-Davis E, Szklo M, Herrington D, Jenny NS, Kronmal R, Barr RG. Nut and seed consumption and inflammatory markers in the multi-ethnic study of atherosclerosis. Am J Epidemiol. 2006 Feb 1;163(3):222-31. doi: 10.1093/aje/kwj033. Epub 2005 Dec 15. PMID 16357111
- See also: Multi Ethnic Study of Atherosclerosis - MESA — http://www.mesa-nhlbi.org